CLINICAL TRIAL: NCT03835234
Title: Incidence of and Factors Associated With Post-operative Nausea and Vomiting Following Surgery Under Regional Anaesthesia
Brief Title: Incidence and Factors Associated With PONV in Regional Anaesthesia
Status: Completed | Type: Observational
Sponsor: Makerere University (Other)
Responsible Party: Sponsor
Other Study IDs: PONVRA
Record Dates: First submitted 2018-09-11; First posted 2019-02-08 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: PONV; Regional Anaesthesia
Keywords: PONV; Regional anaesthesia; LMIC
MeSH Terms: conditions — Postoperative Nausea and Vomiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Post-operative nausea and vomiting (PONV) is one of the complications associated with surgery and anaesthesia. The main aim of the study is to determine the incidence of post-operative nausea and vomiting among surgical patients undergoing regional anaesthesia and the factors associated with it. Patients above the age of 18 who have consented and are undergoing surgery under regional anaesthesia will be enrolled into the study over 6months. They will then be observed for up to 24 hours post operatively to determine the incidence of PONV and factors associated with it.

DETAILED DESCRIPTION:
Post-operative nausea and vomiting (PONV) is one of the complications associated with surgery and anaesthesia. Due to advanced techniques in the field of anaesthesia and surgery, patients are commonly operated on under regional anaesthesia (RA) rather than general anaesthesia (GA). Post-operative nausea and vomiting (PONV) still occurs with regional anaesthesia, but the incidence and associated factors in our setting remain unknown. An optimal management of PONV is important because they can lead to increased morbidity.

The main aim of the study is to determine the incidence of post-operative nausea and vomiting among surgical patients undergoing regional anaesthesia and the factors associated with it.

This will be a prospective cohort study. Patients aged 18 years and above in whom surgery under regional anaesthesia is planned at Mulago hospital will be consented and enrolled into the study over 6months. Data will be collected using semi structured and pre-tested questionnaires. Patients will be observed for up to 24 hours post operatively to determine the incidence of and factors associated with PONV in regional anaesthesia at Mulago hospital. After recruitment, patients will be followed up once at 24 hours post-operatively.

Results from this study will determine the incidence of post-operative nausea and vomiting in surgical patients undergoing regional anaesthesia and the associated factors, data which we do not have in our setting. This will help to guide practice on the prevention and management of post-operative nausea and vomiting.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing regional anaesthesia for emergency or elective surgery.
* Patients aged 18 years and above.
* ASA class 1, 2, 3 and 4 patients

Exclusion Criteria:

* Patients who are switched to general anaesthesia after planned regional anaesthesia.
* Patients with pre-existing nausea and vomiting from co-morbidities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The target populations are all patients 18 years of age and above scheduled for an elective or emergency surgical procedure under regional anaesthesia at Mulago hospital.
  The accessible population includes all patients attending Mulago hospital for elective and emergency surgery under regional anaesthesia during the study period.
Sampling Method: Probability Sample
Enrollment: 364 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
incidence of post operative nausea and vomiting following surgery under regional anaesthesia at Mulago hospital | 24 hours
  Any retching, nausea or vomiting within 24 hours following surgery under regional anaesthesia in Mulago hospital
factors associated with post operative nausea and vomiting following surgery under anaesthesia at Mulago hospital using the Apfel score. | 24 hours
  to determine factors associated with post operative nausea and vomiting following surgery under regional anaesthesia at Mulago hospital using the Apfel score.
  The Apfel score is a verified risk score for predicting post operative nausea and vomiting.It describes four risk factors that when present are scored 1 point each and 0 points when absent. These four risk factors are: use of post operative opioids, female gender, non-smoking status and history of post operative nausea and vomiting or motion sickness. The highest possible score is 4 and lowest possible score is 0.

SECONDARY OUTCOMES:
Proportion of patients that received prophylaxis against post operative nausea and vomiting during surgery under regional anaesthesia at Mulago hospital | 24 hours
  Proportion of patients who received prophylaxis against post operative nausea and vomiting during surgery under regional anaesthesia at Mulago hospital

CONTACTS AND LOCATIONS:
Overall Officials: Dorothy Turitwenka, Principal Investigator — Makerere University
Locations (1):
- Mulago hospital, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (3):
  • Study Protocol (2019-01-31): https://cdn.clinicaltrials.gov/large-docs/34/NCT03835234/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-31): https://cdn.clinicaltrials.gov/large-docs/34/NCT03835234/SAP_001.pdf
  • Informed Consent Form (2018-08-01): https://cdn.clinicaltrials.gov/large-docs/34/NCT03835234/ICF_002.pdf